CLINICAL TRIAL: NCT03045705
Title: Evaluation of the Effect the Medical Team in the Delivery Room Has on Pain Management During Labor.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problem with patient recruitment
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Primary investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0071-17-RMB
Record Dates: First submitted 2017-02-05; First posted 2017-02-07 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Labor Pain
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Labor+routine pain management (Active Comparator): Women that will be treated by the medical team in the delivery room as if not part of a study regarding pain management.
  Interventions: Behavioral: Routine pain management
- Labor+experimental pain management (Active Comparator): Women that will not be asked at all by the medical team in the delivery room regarding analgesia during labor but will be able to receive analgesia at wish at the time of choice.
  Interventions: Behavioral: No inquiry regarding analgesia

INTERVENTIONS:
Behavioral: Routine pain management — Women that will be asked according to the routine management regarding pain management during labor, meaning frequent inquiries regarding the woman's wishes to receive analgesia by the medical team.
  Arms: Labor+routine pain management
Behavioral: No inquiry regarding analgesia — women will not be asked about analgesia during labor by the medical team, but will be able to receive the modality of choice at the time of choice.
  Arms: Labor+experimental pain management

SUMMARY:
In the current study the investigators wish to evaluate the effect the doctors and midwives in the delivery room have on the timing and modality of analgesia chosen by the participants. The participants will be randomly divided into 2 groups. Both groups will be advised of the different modalities of analgesia available during labor. One group will be managed in the delivery room the same as if not part of the study, meaning the doctors and midwives will treat the participants the way they usually do regarding analgesia. The second group of participants will not be asked by the doctors and midwives about analgesia at all but will be able to receive analgesia by a modality of choice at the timing of choice.

DETAILED DESCRIPTION:
After explaining to the participants the study and having signed a confirmed consent, participants will receive an extensive explanation regarding the different modalities of analgesia available during labor. After the explanations the participants will be randomly divided into 2 groups:

1. Routine management-doctors and midwives will treat the participants the way they usually do regarding analgesia including frequent inquiries about wishes for analgesia.
2. Interventional management-participants will not be asked by the doctors and midwives about analgesia at all during labor but will be able to receive analgesia by a modality of choice at the timing of choice after being advised by the medical team.

After delivery, participants will fill a questionnaire regarding the experience of labor in general and the relevance of analgesia during labor including the effect the medical team may have had on decision making during labor.

Medical information regarding visual analogue scale (VAS), analgesia modality, cervical conditions, parity etc. will be extracted from patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Women planned for vaginal delivery.

Exclusion Criteria:

* Women planned for cesarean section.
* Women with comorbidities related to pain that may exacerbate during labor.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale at the time of epidural anesthesia | Up to 3 days from admission.
  Visual analogue scale as reflected by the participant at the time of choice to receive epidural anesthesia.

SECONDARY OUTCOMES:
Visual analogue scale at the time of first medical analgesia | Up to 3 days from admission.
  Visual analogue scale as reflected by the participant at the time of choice to receive the first modality of analgesia.
Analgesia during labor | Up to 3 days from admission.
  Which modalities of analgesia the participant took during labor
Cervical dilatation at the time of epidural anesthesia | Up to 3 days from admission.
  Cervical dilatation at the time of choice to receive epidural anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No